CLINICAL TRIAL: NCT03631329
Title: Predictability of Preoperative Carotid Artery Corrected Flow Time for Hypotension After Spinal Anesthesia in Patients Undergoing Cesarean Section
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0594
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-05

CONDITIONS: Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uncomplicated cesarean delivery: Uncomplicated singleton full-term parturients undergoing cesarean delivery
  Interventions: Diagnostic Test: Doppler sonographic measurement

INTERVENTIONS:
Diagnostic Test: Doppler sonographic measurement — First, place a 4.5-12.0 MHz linear array transducer vertically on the neck with the probe marker facing the patient's head. A long axis B-mode image of the right common carotid artery is obtained at the lower border of the thyroid cartilage. The sample volume is then placed in the center of the lumen located approximately 2 cm proximal to the carotid bifurcation. Next, pulsed wave Doppler tracing is performed in the arterial blood flow. The cycle time using the calliper function in an ultrasonic machine is obtained by measuring the interval between heartbeats at the beginning of the Doppler blood flow upstroke and the Flow time is measured as the time from the beginning of the systolic upstroke to the dicrotic notch.

SUMMARY:
The purpose of this study was to investigate the incidence of hypotension after spinal anesthesia in patients undergoing cesarean section as predicted by preoperative carotid artery corrected flow time measured by Doppler ultrasound. Before entering the operation room, Two inspectors perform two measurements of carotid artery corrected blood flow time respectively, and an average of the four measurements is calculated and analyzed. At this time, the patient's posture is supine, and the head is turned about 30 degrees to the left. Corrected blood flow time (FTc) is measured using carotid ultrasound as previously described by Blehar and colleagues. Corrected blood flow time is calculated by Bazett's formular and Wodey's formular by evaluating a single cycle after several successive cycles have reached a stable and acceptable quality level.

The occurrence of hypotension is recorded from the spinal anesthetic injection until the fetus is delivered.

The definition of hypotension after spinal anesthesia is that the systolic blood pressure drops to 80 mmHg, less than 75% of the baseline value, or even if it does not meet the former criteria, symptoms that are consistent with hypotension (dizziness, dizziness, dyspnea, nausea or vomiting).

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated singleton full-term parturients undergoing cesarean delivery
* age 20~40
* ASA class 1~3

Exclusion Criteria:

* Emergency surgery
* Placenta previa
* Preeclampsia or Preeclampsia
* Cardiovascular or cerebrovascular disease
* Morbid obesity with a body mass index (BMI) of 40 kg / m2 or higher
* Gestational age <36 or ≥ 41 weeks
* Contraindications to spinal anesthesia
* Carotid stenosis> 50% (angiography, CT angiography, MR angiography, or duplex ultrasonography)
* Basal systolic blood pressure> 160 mmHg
* The preoperative examination revealed that the electrocardiogram was not normal sinus rhythm
* Chronic kidney disease (eGFR <60 mL / min / 1.73 m2)
* If the subject includes a person who can not read the written consent (eg, illiterate, foreigner, etc.)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Uncomplicated singleton full-term parturients undergoing cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of Hypotension | from the spinal anesthetic injection until the fetus is delivered.
  The definition of hypotension after spinal anesthesia is that the systolic blood pressure drops to 80 mmHg, less than 75% of the baseline value , or even if it does not meet the former criteria, symptoms that are consistent with hypotension (dizziness, dizziness, dyspnea, nausea or vomiting) .

SECONDARY OUTCOMES:
The systolic blood pressure difference | from the spinal anesthetic injection until the fetus is delivered.
  The most significant difference in systolic blood pressure dropped

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HJ, Choi YS, Kim SH, Lee W, Kwon JY, Kim DH. Predictability of preoperative carotid artery-corrected flow time for hypotension after spinal anaesthesia in patients undergoing caesarean section: A prospective observational study. Eur J Anaesthesiol. 2021 Apr 1;38(4):394-401. doi: 10.1097/EJA.0000000000001376. PMID 33122575